CLINICAL TRIAL: NCT03959267
Title: Testing a Culturally Adapted Telephone Genetic Counseling Intervention to Enhance Genetic Risk Assessment in Underserved Latinas at Risk of Hereditary Breast and Ovarian Cancer
Brief Title: Testing a Culturally Adapted Telephone Genetic Counseling Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Hackensack Meridian Health (Other)
Responsible Party: Principal Investigator, Alejandra Hurtado de Mendoza, Assistant Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KL2TR001432 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-22 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer; Hereditary Breast Cancer
Keywords: Latinas; Survivors
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer, Familial

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a two-arm Randomized Controlled Trial (RCT) comparing Telephone Genetic Counseling in Spanish vs. Usual care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will continue with their usual medical care. Usual care may vary at different sites. Based on the investigator's preliminary data usual care can result in not GCRA referral, referral directly to testing, or referral to genetic counseling with an interpreter. The investigators will document usual care for participants from the sites randomized to usual care.
- Telephone Genetic Counseling (Other): Participants will receive telephone genetic counseling with the culturally adapted protocol and booklet
  Interventions: Behavioral: Telephone Genetic Counseling

INTERVENTIONS:
Behavioral: Telephone Genetic Counseling — A genetic counselor fluent in Spanish (see letter of support) will conduct the TGC. The TGC intervention consists of two sessions. Prior to the sessions the investigators will mail participants the education materials with information to be reviewed prior to the genetic counseling session and a set of visual aids that the counselor will refer to during the session to facilitate the understanding of the information conveyed in the session.
  Arms: Telephone Genetic Counseling

SUMMARY:
Participating in genetic cancer risk assessments (GCRA) for hereditary breast and ovarian cancer (HBOC) can inform treatment and risk management decisions and improve breast cancer outcomes. However, Latina women underuse GCRA services, which may increase breast cancer disparities. This study will adapt and test the impact of a Culturally Adapted Telephone Genetic Counseling Intervention to enhance the use and quality of genetic counseling services for underserved Latina women at-risk of hereditary breast and ovarian cancer

DETAILED DESCRIPTION:
SPECIFIC AIMS Women with BRCA1/2 mutations have a 50-80% and 15-40% lifetime risk of developing breast and ovarian cancer, respectively.1 Breast cancer survivors with BRCA1/2 mutations are three times more likely to develop contralateral breast cancer than non-carriers.2 The National Comprehensive Cancer Network (NCCN) recommends referral for hereditary breast and ovarian cancer (HBOC) genetic cancer risk assessments (genetic counseling and consideration of genetic testing; GCRA) for women at high risk of carrying a mutation.3 A positive genetic test can inform treatment in newly diagnosed breast cancer patients and management in survivors and unaffected women.4 Latinas have a significantly higher BRCA1/2 gene mutation prevalence than non-Latina Whites,5 yet they are 4-5 times less likely to have GCRA.6 Reasons for lower GCRA use include access, language barriers, and psychosocial factors.7-12 Fewer than 5% of the already limited number of genetic counselors in the US speak a language other than English.13 Developing alternative strategies to enhance GCRA access is important to ensure national guidelines are met and to reduce disparities.5,14

Our preliminary data suggest that GCRA referral guidelines are not consistently met among high-risk Latinas, many of whom are often not offered GCRA or are offered testing without counseling due to access and language barriers. Alternative strategies for delivery of genetic services, such as telephone genetic counseling (TGC), are safe, acceptable, and effective in both urban and rural populations.15,16 TGC can be a viable alternative strategy to in-person counseling for Latinas given that (1) TGC can enhance access to comprehensive genetic counseling by reducing cost and logistic barriers, which are especially important in underserved groups17; (2) TGC can also maximize the reach and access to the few Spanish-speaking genetic counselors in the US.13 Our initial data indicate that providers will increase the number of referrals to GCRA if Spanish genetic counseling is available. Thus, by overcoming access and language barriers, Spanish TGC can increase GCRA access among this high-risk yet underserved population.

Beyond addressing access and language barriers, Spanish TGC may enhance the quality of information conveyed during counseling. Given the shortage of Spanish-speaking genetics professionals, English-speaking counselors use phone or in-person interpretation services with Spanish-speaking patients. Unfortunately, the quality of the information conveyed via Spanish interpreters is suboptimal.18 Interpreters do not have the requisite genetics expertise and may reduce, omit, or revise content.19 An initial study found that during HBOC genetic counseling, interpreters translated probabilistic statements as definitive or shortened and altered key explanations of risk information.18 In addition to potential content inaccuracies, interpretation typically precludes 'small talk' that helps build rapport.20 Our preliminary data align, suggesting both Latinas and providers report concerns about accuracy and rapport in sessions with interpreters. Spanish TGC could improve counseling quality by eliminating the need for interpretation for Latinas who are referred to and attend counseling.

The investigators will compare evidence-based TCG developed by members of my mentoring team16,21 to usual care (UC) among high-risk, Spanish-speaking Latinas. The investigators anticipate that usual care will consist of either no referral to GCRA, offer of direct genetic testing without counseling, or genetic counseling with interpretation. Guided by the Ottawa Framework for Informed Decision Making22 the investigators propose a two phased mixed methods study. In Phase I, the investigators will conduct interviews with high-risk Latinas (n=15) to adapt the intervention materials using the Learner Verification and Revision frame.23 In Phase II, the investigators will use a cluster randomized design with four sites randomized to Spanish TGC (n=2 sites) or UC (n=2 sites). Our primary outcome is genetic counseling uptake among 60 high risk Latinas. Genetic testing uptake will be a secondary outcome. Among women who receive genetic counseling either through TGC or with an interpreter, the investigators will assess counseling quality by evaluating women's knowledge, counseling satisfaction, and communication in 20 audiotaped sessions. The investigators will assess communication using the gold standard RIAS quantitative coding system 24 and qualitative discourse analysis.25 Participants will complete assessments at baseline, post-counseling, and at 3 months. The investigators aim to:

Aim 1. Culturally adapt the TGC booklet and genetic counseling protocols. Aim 2. Evaluate the impact of TGC vs. UC on GCRA access. Participants randomized to TGC (vs. UC) will have H.2.1. higher genetic counseling uptake H.2.2. higher testing uptake 3 months post intervention.

Aim 3. Assess the quality of genetic counseling sessions among participants who attend the sessions. H.3.1. Participants randomized to TGC (vs. UC) will have higher HBOC knowledge and satisfaction and lower decisional conflict and distress. H.3.2. The investigators will explore communication patterns in 20 TGC and genetic counseling sessions with an interpreter using quantitative and qualitative methods.

Given access barriers and the shortage of Spanish speaking genetic counselors, adapting and translating TGC intervention is a promising strategy that could reduce disparities by broadening the reach and accessibility to genetic counseling while enhancing the quality of the service.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Latina/Hispanic
* Be 21 years old or older
* Be at risk of hereditary breast and ovarian cancer because of personal and/or family medical history according to NCCN guidelines
* Be diagnosed with breast cancer, and have completed active treatment (i.e., chemotherapy, radiation, surgeries)
* Be able to provide the name and contact information of a primary healthcare provider, whom they see at least once a year
* Speak and read Spanish.

Exclusion Criteria:

* Do not identify as Latina/Hispanic.
* Younger than 21 years old.
* Do not meet current national guidelines to be considered at risk for hereditary breast and ovarian cancer.
* Has been diagnosed with ovarian cancer or stage IV breast cancer.
* Has not completed active treatment (e.g., surgery, chemotherapy, radiation).
* Is not able to provide the name and contact information of the primary healthcare provider. This must be someone whom they have seen at least once during the past 12 months.
* Cannot provide consent to participate.
* Has received genetic counseling by a genetics professional (e.g., genetic counselor or genetics nurse).
* Has participated in a previous phase of this study.
* Cannot provide a copy of their genetic test results.

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on the self-representation of gender identity
Enrollment: 37 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Number of participants that receive genetic cancer risk assessment (GCRA) | Three months after baseline
  The RA will conduct a follow-up call to inquire whether participants randomized to Usual Care completed a GCRA appointment and to gather information about the place where the appointment was held and name of the genetic counselor

SECONDARY OUTCOMES:
Change in knowledge | Change from baseline to three months after baseline
  The investigators will measure knowledge with the 13-item Breast Cancer Genetic Knowledge Scale by Erblich et al., 2005 answered in a True/False/Do not know format. Answers are recoded to correct or incorrect. The number of correct responses are added to create a score ranging from 0-13. Higher scores mean higher breast cancer genetics knowledge.
Change in decisional conflict | Change from baseline to three months after baseline
  The investigators will measure decisional conflict with the 16-item Decisional-Conflict Scale by O'Connor AM, 1995. The scale is rated on a 1-5 scale. Answers are aggregated to yield a score from 16-80. The higher the final score, the least decisional conflict.
Distress | At baseline
  The investigators will measure distress using the Patient Reported Outcomes Measurement Information System (PROMIS) short anxiety scale by Pilkonis, P.A., Choi, S.W., Reise, S.P., Stover, A.M., Riley, W.T., Cella, D., on behalf of the PROMIS Cooperative Group. (2011). The scale is 1 - 6 scale, in which higher scores mean higher distress.
Decision Satisfaction | Three months after baseline
  The investigators will measure satisfaction with healthcare decisions using the 5 item Satisfaction with healthcare decisions scale by Holmes-Rovner M, Kroll J, Schmitt N, et al., 1996. The scale answers go from 1- 5. The higher scores represent higher satisfaction with healthcare decisions.
Satisfaction with counseling | Three months after baseline
  The investigators use a scale developed by their team, which have been used in prior published work (see DeMarco TA, Peshkin BN, Mars BD, Tercyak KP., 2004 and Tercyak KP, Demarco TA, Mars BD, Peshkin BN., 2004). This 5-item scale is answered from 1-5, with higher scores signifying higher satisfaction with counseling.
Number of participants that receive genetic testing | Three months after baseline
  The RA will conduct a follow-up call to inquire whether participants pursued genetic testing or not.

OTHER OUTCOMES:
Communication | Three months after baseline
  Communication outcomes will be qualitatively measured using discourse analysis (e.g., "Number of patient-initiated questions" will be coded following guidelines).
Communication | Three months after baseline
  Communication outcomes will be quantitatively measured following RIAS medical interaction coding guidelines (e.g., patient centeredness).
Acceptability | Thee months after baseline
  Using a 12-item scale, the RA will assess whether participants perceived the genetic counseling session as acceptable or not based on answers from 1 - 10 and "Strongly disagree" to "Strongly agree"

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Hurtado de Mendoza, PhD, Principal Investigator — Georgetown University
Locations (4):
- United States (4):
  - Capital Breast Care Center, Washington D.C., District of Columbia
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Nueva Vida, Alexandria, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Chen S, Parmigiani G. Meta-analysis of BRCA1 and BRCA2 penetrance. J Clin Oncol. 2007 Apr 10;25(11):1329-33. doi: 10.1200/JCO.2006.09.1066. PMID 17416853
- [Background] Valachis A, Nearchou AD, Lind P. Surgical management of breast cancer in BRCA-mutation carriers: a systematic review and meta-analysis. Breast Cancer Res Treat. 2014 Apr;144(3):443-55. doi: 10.1007/s10549-014-2890-1. Epub 2014 Feb 25. PMID 24567198
- [Background] Kauff ND, Satagopan JM, Robson ME, Scheuer L, Hensley M, Hudis CA, Ellis NA, Boyd J, Borgen PI, Barakat RR, Norton L, Castiel M, Nafa K, Offit K. Risk-reducing salpingo-oophorectomy in women with a BRCA1 or BRCA2 mutation. N Engl J Med. 2002 May 23;346(21):1609-15. doi: 10.1056/NEJMoa020119. Epub 2002 May 20. PMID 12023992
- [Background] Weitzel JN, Clague J, Martir-Negron A, Ogaz R, Herzog J, Ricker C, Jungbluth C, Cina C, Duncan P, Unzeitig G, Saldivar JS, Beattie M, Feldman N, Sand S, Port D, Barragan DI, John EM, Neuhausen SL, Larson GP. Prevalence and type of BRCA mutations in Hispanics undergoing genetic cancer risk assessment in the southwestern United States: a report from the Clinical Cancer Genetics Community Research Network. J Clin Oncol. 2013 Jan 10;31(2):210-6. doi: 10.1200/JCO.2011.41.0027. Epub 2012 Dec 10. PMID 23233716
- [Background] Dean M, Boland J, Yeager M, Im KM, Garland L, Rodriguez-Herrera M, Perez M, Mitchell J, Roberson D, Jones K, Lee HJ, Eggebeen R, Sawitzke J, Bass S, Zhang X, Robles V, Hollis C, Barajas C, Rath E, Arentz C, Figueroa JA, Nguyen DD, Nahleh Z. Addressing health disparities in Hispanic breast cancer: accurate and inexpensive sequencing of BRCA1 and BRCA2. Gigascience. 2015 Nov 4;4:50. doi: 10.1186/s13742-015-0088-z. eCollection 2015. PMID 26543556
- [Background] Glenn BA, Chawla N, Bastani R. Barriers to genetic testing for breast cancer risk among ethnic minority women: an exploratory study. Ethn Dis. 2012 Summer;22(3):267-73. PMID 22870568
- [Background] Sussner KM, Jandorf L, Thompson HS, Valdimarsdottir HB. Barriers and facilitators to BRCA genetic counseling among at-risk Latinas in New York City. Psychooncology. 2013 Jul;22(7):1594-604. doi: 10.1002/pon.3187. Epub 2012 Sep 16. PMID 22987526
- [Background] Sussner KM, Edwards T, Villagra C, Rodriguez MC, Thompson HS, Jandorf L, Valdimarsdottir HB. BRCA genetic counseling among at-risk Latinas in New York City: new beliefs shape new generation. J Genet Couns. 2015 Feb;24(1):134-48. doi: 10.1007/s10897-014-9746-z. Epub 2014 Aug 15. PMID 25120034
- [Background] Sussner KM, Jandorf L, Thompson HS, Valdimarsdottir HB. Interest and beliefs about BRCA genetic counseling among at-risk Latinas in New York City. J Genet Couns. 2010 Jun;19(3):255-68. doi: 10.1007/s10897-010-9282-4. Epub 2010 Feb 12. PMID 20151317
- [Background] Thompson HS, Valdimarsdottir HB, Jandorf L, Redd W. Perceived disadvantages and concerns about abuses of genetic testing for cancer risk: differences across African American, Latina and Caucasian women. Patient Educ Couns. 2003 Nov;51(3):217-27. doi: 10.1016/s0738-3991(02)00219-7. PMID 14630378
- [Background] Armstrong K, Micco E, Carney A, Stopfer J, Putt M. Racial differences in the use of BRCA1/2 testing among women with a family history of breast or ovarian cancer. JAMA. 2005 Apr 13;293(14):1729-36. doi: 10.1001/jama.293.14.1729. PMID 15827311
- [Background] Hall MJ, Olopade OI. Disparities in genetic testing: thinking outside the BRCA box. J Clin Oncol. 2006 May 10;24(14):2197-203. doi: 10.1200/JCO.2006.05.5889. PMID 16682739
- [Background] Schwartz MD, Valdimarsdottir HB, Peshkin BN, Mandelblatt J, Nusbaum R, Huang AT, Chang Y, Graves K, Isaacs C, Wood M, McKinnon W, Garber J, McCormick S, Kinney AY, Luta G, Kelleher S, Leventhal KG, Vegella P, Tong A, King L. Randomized noninferiority trial of telephone versus in-person genetic counseling for hereditary breast and ovarian cancer. J Clin Oncol. 2014 Mar 1;32(7):618-26. doi: 10.1200/JCO.2013.51.3226. Epub 2014 Jan 21. PMID 24449235
- [Background] Kinney AY, Butler KM, Schwartz MD, Mandelblatt JS, Boucher KM, Pappas LM, Gammon A, Kohlmann W, Edwards SL, Stroup AM, Buys SS, Flores KG, Campo RA. Expanding access to BRCA1/2 genetic counseling with telephone delivery: a cluster randomized trial. J Natl Cancer Inst. 2014 Nov 5;106(12):dju328. doi: 10.1093/jnci/dju328. Print 2014 Dec. PMID 25376862
- [Background] Joseph G, Guerra C. To worry or not to worry: breast cancer genetic counseling communication with low-income Latina immigrants. J Community Genet. 2015 Jan;6(1):63-76. doi: 10.1007/s12687-014-0202-4. Epub 2014 Aug 23. PMID 25148879
- [Background] Aranguri C, Davidson B, Ramirez R. Patterns of communication through interpreters: a detailed sociolinguistic analysis. J Gen Intern Med. 2006 Jun;21(6):623-9. doi: 10.1111/j.1525-1497.2006.00451.x. PMID 16808747
- [Background] Browner CH, Preloran HM, Casado MC, Bass HN, Walker AP. Genetic counseling gone awry: miscommunication between prenatal genetic service providers and Mexican-origin clients. Soc Sci Med. 2003 May;56(9):1933-46. doi: 10.1016/s0277-9536(02)00214-9. PMID 12650730
- [Background] O'Connor AM, Stacey D, Rovner D, Holmes-Rovner M, Tetroe J, Llewellyn-Thomas H, Entwistle V, Rostom A, Fiset V, Barry M, Jones J. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2001;(3):CD001431. doi: 10.1002/14651858.CD001431. PMID 11686990
- [Background] Roter D, Larson S. The Roter interaction analysis system (RIAS): utility and flexibility for analysis of medical interactions. Patient Educ Couns. 2002 Apr;46(4):243-51. doi: 10.1016/s0738-3991(02)00012-5. PMID 11932123
- [Background] Kinney AY, Gammon A, Coxworth J, Simonsen SE, Arce-Laretta M. Exploring attitudes, beliefs, and communication preferences of Latino community members regarding BRCA1/2 mutation testing and preventive strategies. Genet Med. 2010 Feb;12(2):105-15. doi: 10.1097/GIM.0b013e3181c9af2d. PMID 20061960
- [Background] Erblich J, Brown K, Kim Y, Valdimarsdottir HB, Livingston BE, Bovbjerg DH. Development and validation of a Breast Cancer Genetic Counseling Knowledge Questionnaire. Patient Educ Couns. 2005 Feb;56(2):182-91. doi: 10.1016/j.pec.2004.02.007. PMID 15653247
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Horowitz M, Wilner N, Alvarez W. Impact of Event Scale: a measure of subjective stress. Psychosom Med. 1979 May;41(3):209-18. doi: 10.1097/00006842-197905000-00004. PMID 472086
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600
- [Background] DeMarco TA, Peshkin BN, Mars BD, Tercyak KP. Patient satisfaction with cancer genetic counseling: a psychometric analysis of the Genetic Counseling Satisfaction Scale. J Genet Couns. 2004 Aug;13(4):293-304. doi: 10.1023/b:jogc.0000035523.96133.bc. PMID 19736695
- [Background] Tercyak KP, Demarco TA, Mars BD, Peshkin BN. Women's satisfaction with genetic counseling for hereditary breast-ovarian cancer: psychological aspects. Am J Med Genet A. 2004 Nov 15;131(1):36-41. doi: 10.1002/ajmg.a.30317. PMID 15389697
- [Derived] Gomez-Trillos S, Graves KD, Fiallos K, Schwartz MD, Peshkin BN, Hamilton H, Sheppard VB, Vadaparampil ST, Campos C, Cupertino AP, Alzamora MC, Lynce F, Hurtado-de-Mendoza A. Cultural adaptations to a telephone genetic counseling protocol and booklet for Latina breast cancer survivors at risk for hereditary breast and ovarian cancer. Transl Behav Med. 2023 May 13;13(5):297-308. doi: 10.1093/tbm/ibac106. PMID 36694918